CLINICAL TRIAL: NCT04644471
Title: Comparison Between Ultra-low-dose Computed Tomography and Lung MRI for Morphological Assessment of Lung Disease in Adult Cystic Fibrosis Patients
Brief Title: Comparison Between Ultra-low-dose Computed Tomography and Lung MRI in Cystic Fibrosis
Acronym: UBD-IRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP190061; 2019-A02078-49 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-10-05; First posted 2020-11-25 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Cystic Fibrosis
Keywords: Magnetic resonance imaging; Multidetector computed tomography
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: CT scanner — 1 conventional low dose inspiratory acquisition and 1 ultra-low-dose inspiratory acquisition
Diagnostic Test: Lung MRI — 3 UTE sequences (free breathing, inspiratory and expiratory) and 1 T2 sequence

SUMMARY:
The purpose of this study is to compare the performances of ultra-low dose computed tomography (CT) and lung magnetic resonance imaging (MRI) for morphological assessment of cystic fibrosis-related lung disease and to compare their performances to conventional low dose CT

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a recessive autosomal disease caused by mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene that encodes for an epithelial chloride channel involved in ion and fluid transport. CF is the most common inherited disease in Caucasians and disease severity mainly depends on the degree of lung involvement, which can lead to terminal respiratory failure Disease monitoring of CF-related lung disease rely on functional assessment and complimentary morphological assessment. Conventional low-dose chest computed tomography (CT) is currently the gold standard for the morphological assessment of CF-related lung disease but ultra-low dose chest CT and high-resolution magnetic resonance imaging (MRI) of the lung using UTE sequences have been recently developed and allow important radiation reduction of radiation dose exposure. However the performances of these 2 competing imaging methods remains to be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year-old
* Diagnosis of cystic fibrosis provided by genetic and swear test
* Chest CT acquisition performed as part of the standard follow-up
* Patient with social security or health insurance
* Informed consent

Exclusion Criteria:

* MRI contraindication
* Orthopnea
* Inability to hold breath for 17 seconds
* No spirometry planned the same day
* Lung transplant patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Reproducibility of visual score between imaging modalities | 1 day
  Reproducibility disease severity measured by the Helbich scoring system with conventional CT as gold standard

SECONDARY OUTCOMES:
Intra and interobserver reproducibility of visual scores | 1 day
  Intra and interobserver reproducibility of the Helbich score for each imaging modality
Correlation between visual scores and pulmonary function | 1 day
  Correlation between the Helbich score for each imaging modality and forced expiratory volume in 1 second (FEV1)
Correlation between air trapping at MRI and pulmonary function test | 1 day
  Correlation between air trapping, measured by comparing inspiratory to expiratory MRI images, and forced expiratory volume at one second (FEV1)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre REVEL, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dournes G, Grodzki D, Macey J, Girodet PO, Fayon M, Chateil JF, Montaudon M, Berger P, Laurent F. Quiet Submillimeter MR Imaging of the Lung Is Feasible with a PETRA Sequence at 1.5 T. Radiology. 2015 Jul;276(1):258-65. doi: 10.1148/radiol.15141655. Epub 2015 Mar 13. PMID 25768672
- [Background] Dournes G, Menut F, Macey J, Fayon M, Chateil JF, Salel M, Corneloup O, Montaudon M, Berger P, Laurent F. Lung morphology assessment of cystic fibrosis using MRI with ultra-short echo time at submillimeter spatial resolution. Eur Radiol. 2016 Nov;26(11):3811-3820. doi: 10.1007/s00330-016-4218-5. Epub 2016 Feb 2. PMID 26843010
- [Background] Chassagnon G, Martin C, Ben Hassen W, Freche G, Bennani S, Morel B, Revel MP. High-resolution lung MRI with Ultrashort-TE: 1.5 or 3 Tesla? Magn Reson Imaging. 2019 Sep;61:97-103. doi: 10.1016/j.mri.2019.04.015. Epub 2019 Apr 30. PMID 31051201
- [Background] Chassagnon G, Martin C, Marini R, Vakalopolou M, Regent A, Mouthon L, Paragios N, Revel MP. Use of Elastic Registration in Pulmonary MRI for the Assessment of Pulmonary Fibrosis in Patients with Systemic Sclerosis. Radiology. 2019 May;291(2):487-492. doi: 10.1148/radiol.2019182099. Epub 2019 Mar 5. PMID 30835186